CLINICAL TRIAL: NCT04407767
Title: Personalizing Cognitive Processing Therapy With a Case Formulation Approach to Intentionally Target Impairment in Psychosocial Functioning Associated With PTSD
Brief Title: A Case Formulation Approach to Cognitive Processing Therapy
Acronym: CF-CPT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F3369-R
Record Dates: First submitted 2020-05-08; First posted 2020-05-29 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Cognitive Processing Therapy; Case Formulation; Functional Outcomes; Psychosocial Functioning
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This randomized controlled clinical trial seeks to examine the relative efficacy of a case formulation approach integrated into cognitive processing therapy as compared to standard cognitive processing therapy. Randomization to study condition will occur at the provider level (50 providers will be randomized to either CPT or CF-CPT. Each provider will treat the next 4 eligible veterans (total sample = 200 Veterans) seeking care for PTSD who agree to participate in the study.
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators will be blind to treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case Formulation plus Cognitive Processing Therapy (Experimental): The CF approach alters the CPT protocol in two ways: expanding the protocol to intentionally and systematically address impairment in functioning, and enhancing the providers' latitude to navigate challenges to optimal therapy outcomes (COTOS). CF-CPT begins with a formal CF assessment session; elements of CF are then integrated throughout CPT. CF modifications to the original CPT protocol occur in each session by intentionally attending to cognitions that are impeding the patient's functional recovery. The second modification includes enhancing the provider's latitude to diverge from the protocol when clinically wise. CF-CPT provides guidance around the identification, monitoring and management of COTOs, and, importantly, the expedient return to the CPT protocol with continued attention to COTOs.
  Interventions: Behavioral: Case Formulation plus Cognitive Processing Therapy
- Cognitive Processing Therapy (Active Comparator): CPT is a brief therapy for PTSD predominantly based on cognitive theory. Traditionally delivered over 12 one-hour sessions weekly or twice weekly, CPT is now variable length depending on patient's recovery from PTSD. CPT is delivered in three phases: education, processing, and challenging and focuses on challenging beliefs and assumptions related to the trauma, oneself, and the world. Changing dysfunctional beliefs alters negative emotions emanating from those beliefs.
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Case Formulation plus Cognitive Processing Therapy — The CF approach alters the CPT protocol in two ways: expanding the protocol to intentionally and systematically address impairment in functioning, and enhancing the providers' latitude to navigate challenges to optimal therapy outcomes (COTOS). CF-CPT begins with a formal CF assessment session; elements of CF are then integrated throughout CPT. CF modifications to the original CPT protocol occur in each session by intentionally attending to cognitions that are impeding the patient's functional recovery. The second modification includes enhancing the provider's latitude to diverge from the protocol when clinically wise. CF-CPT provides guidance around the identification, monitoring and management of COTOs, and, importantly, the expedient return to the CPT protocol with continued attention to COTOs.
  Arms: Case Formulation plus Cognitive Processing Therapy
Behavioral: Cognitive Processing Therapy — CPT is a brief therapy for PTSD predominantly based on cognitive theory. Traditionally delivered over 12 one-hour sessions weekly or twice weekly, CPT is now variable length depending on patient's recovery from PTSD. CPT is delivered in three phases: education, processing, and challenging and focuses on challenging beliefs and assumptions related to the trauma, oneself, and the world. Changing dysfunctional beliefs alters negative emotions emanating from those beliefs.
  Arms: Cognitive Processing Therapy

SUMMARY:
Recent estimates suggest that over 610,000 US Veterans treated by the Veterans Health Administration (VHA) suffer from PTSD, a disorder that can be chronic and debilitating. The heterogeneity of the 20 symptoms of PTSD; comorbidity with disorders such as depression, panic, and substance use; high rates of lingering effects of physical injury; and suicidality all contribute to complex clinical presentations and can exact a significant toll on functioning, quality of life, and well-being even decades after exposure to the traumatic event. Perhaps spurred by the President's New Freedom Commission on Mental Health, psychosocial rehabilitation has shifted from the periphery in mental health recovery models to a more primary focus in clinical settings, including recommendations for use of psychosocial rehabilitation techniques in trauma-focused mental health care. Support for the efficacy of psychosocial rehabilitation techniques in PTSD recovery programs has burgeoned in recent years and data supporting psychological treatments for PTSD has increased exponentially, yet the two approaches to recovery have largely remained independent.

Cognitive Processing Therapy (CPT), the evidence-based psychotherapy (EBP) for PTSD most frequently delivered within VHA, yields large magnitude reductions in primary PTSD outcomes. Corresponding gains in occupational, social, leisure, and sexual functioning, and in health-related concerns have also been demonstrated. Despite CPT's effectiveness, there is room for improvement in overall outcomes and patient engagement. Further, improvements in functioning and quality of life are more modest than those observed in PTSD and associated mental health symptoms. Prior work suggests that unaddressed difficulties in functioning contribute to premature dropout from EBPs for PTSD among Veterans. Directly targeting impairments associated with psychosocial functioning has the potential to substantially increase the scope of recovery beyond the core symptoms of PTSD and facilitate greater patient engagement, resulting in more Veterans benefitting from CPT. Modifying the CPT protocol to personalize the intervention for the individual patient has resulted in better overall response rates for a wider variety of patient populations suffering from complicated clinical presentations.

Case formulation (CF) is a well-established approach to cognitive-behavioral treatment that facilitates a collaborative process between providers and patients to guide the tailoring of treatment to meet idiosyncratic patient needs. Integrating CF strategies into the existing CPT protocol will enable providers to personalize CPT to directly address impairment in functioning as well as provide the latitude to directly intervene with the complex challenges that threaten optimal outcomes within the context of trauma-focused therapy. CF-integrated CPT (CF-CPT) expands and enhances the CPT protocol to facilitate a personalized and flexible approach to treating PTSD that prioritizes the administration of the full dose of CPT while expanding the protocol to directly target important domains of functioning and result in more holistic outcomes.

This controlled treatment outcome trial will randomize a national sample of CPT providers (Veteran n = 200; provider n = 50) to either deliver CF-CPT or CPT to compare the relative effectiveness of CF-CPT to CPT in improving primary outcomes, including Veterans' psychosocial functioning, quality of life and well-being over the course of treatment and 3-month follow-up as compared to Veterans who receive standard CPT. Further, Veterans who receive CF-CPT will demonstrate greater reductions in PTSD and depression over the course of treatment and 3-month follow-up than those who receive CPT.

This study also seeks to determine the effectiveness of CF-CPT as compared to CPT in improving Veterans' treatment engagement (CF-CPT will demonstrate higher rates of Veteran treatment completion than CPT).

This study will valuate CF-CPT's indirect impact on Veterans' psychosocial functioning and PTSD/depression symptomology Change in functioning, quality of life, and well-being & PTSD and depression will be associated with improvement in the idiosyncratic clinical challenges targeted by the CF.

This study will also examine between-group differences across secondary outcomes (e.g. anger, anxiety, health concerns, sleep, numbing/reactivity) and describe the frequency and type of the clinical and rehabilitative needs of the Veterans and the type and duration of divergences (e.g. rehabilitative techniques) made by providers.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is common and complicated. Recent estimates suggest that over 610,000 US Veterans treated by the Veterans Health Administration (VHA) suffer from posttraumatic stress disorder (PTSD), a disorder that can be chronic and debilitating. The heterogeneity of the 20 symptoms of PTSD; comorbidity with disorders such as depression, panic, and substance use; high rates of concurrent and lingering effects of physical injury, and suicidality all contribute to complex clinical presentations and can exact a significant toll on functioning, quality of life, and well-being decades after exposure to the trauma. The complex and enduring challenges inherent in PTSD and their effect on patients' functioning pose significant hurdles for patients and clinicians.

Impairments in psychosocial functioning are an important, but less well-attended, facet of PTSD. While significant impairment in functioning is clearly a requirement for the diagnosis of PTSD as indicated by Criterion G of the diagnostic criteria for PTSD, resolution of functional impairment is not considered to be a primary therapeutic target in evidence-based PTSD treatment protocols. Improvements in domains of functioning and, more broadly, quality of life and well-being, are most typically considered secondary outcomes in RCTs, if they are reported at all. This seeming lack of attention to impairments in functioning stands in stark contrast to patients' reports of the meaningfulness of these impairments in their lives. In fact, it is often precisely these types of impairments that drive patients suffering from PTSD to seek treatment, arguably more so than the 20 core symptoms of the disorder.

Researchers and providers alike recognize the importance of well-being and seek to maximize functional recovery. It has theoretically been difficult to directly target impairment in functioning (PTSD Criterion G) in manualized therapies, perhaps because "functional impairment" is quite variable across patients in breadth and scope. Including explicit and manualized instruction on "treating functional impairment" is impossible and is likely the reason that no single PTSD psychotherapy exists that is specifically designed to "treat" functional recovery. Trauma-focused EBPs instead are specifically designed to directly target the core symptoms of PTSD. Functional impairment is targeted indirectly through relief in the core symptoms. For example, improvement in occupational functioning may be achieved through decreases in avoidance, mood or anger symptoms that might be interfering with job performance. Gains in functioning (e.g. improving marital relations or workplace functioning) and large effects in well-being and quality of life have historically been difficult to operationalize and are often considered more longterm therapeutic goals, perhaps beyond the scope of brief therapies. However, given the importance of functioning to patients with PTSD, intentionally and thoughtfully building on the success of the skills acquired in evidence-based psychotherapies (EBPs) and expanding those skills to specifically target functional outcomes warrants further exploration.

Cognitive Processing Therapy (CPT) is effective at reducing PTSD symptoms and is widely used. CPT is one of the therapies with the most accumulated empirical support to date. Recent meta-analyses indicate that CPT has the largest effect size of existing evidence-based treatments for PTSD in soldiers and Veterans and across trauma populations (mean ES = 1.69). The effectiveness of CPT extends across patient populations suffering from a range of comorbid conditions including TBI, chronic child abuse histories, comorbid psychiatric and substance use disorders, and ongoing peritraumatic situations. CPT has been designated a first-line treatment in a number of clinical guidelines, including the VHA / Department of Defense (DoD) PTSD Clinical Practice Guidelines. Since 2007, VHA has dedicated substantial resources and effort to the historic, large-scale dissemination of CPT via the Mental Health Dissemination Initiative. To date, over 4,150 VHA providers have been trained in CPT and at least 20,774 Veterans have begun CPT in the last year. Yet the impact of CPT on both PTSD symptoms and psychosocial functioning can be improved.

Veterans with PTSD present to treatment with challenges in psychosocial functioning and other clinical complexities; the failure of manualized treatments for PTSD to provide guidance on how to address these concerns is negatively impacting outcomes. Nearly all (87%) Veterans with PTSD presenting to VHA primary care have at least one comorbid psychiatric condition and, on average, Veterans with PTSD had 2.95 comorbid mental health diagnoses and over 50% reported suicidal ideation. Across trauma populations, PTSD is associated with severe impairments in social and occupational functioning, exerting a more deleterious effect than most mental health diagnoses. Clinical presentations in Veterans suffering from PTSD are further complicated by a host of psychosocial stressors, impairments in major domains of functioning, and comorbid physical conditions. Veterans are more likely to be homeless, be under- or unemployed, and have poor physical health status as compared to non-Veterans. Prior work suggests that unaddressed difficulties in these domains contributes to suboptimal outcomes and premature dropout from CPT among Veterans. The investigators posit that frontline treatments for PTSD must be expanded to directly and intentionally target functional impairments and improve holistic outcomes.

While fidelity to the CPT protocol is essential, skillful divergences can be clinically wise. Administering EBPs in a standardized manner is critical to ensuring that patients receive an accurate and adequate dose of the intervention. Yet, as outlined above, strict protocol adherence (e.g., failing to assess and address psychosocial stressors and other clinical complexities) may result in premature abandonment of trauma-focused therapy and/or suboptimal outcomes. Modifications to the CPT protocol can enhance therapy outcomes. The next step in this program of research is to leverage the success of CPT in treating core symptoms of PTSD and expand the protocol to directly target functional outcomes. Thoughtfully and intentionally enhancing the latitude of the CPT protocol to target clinical complexities that pose a risk to holistic outcomes personalizes the delivery of care to best meet the individual patient's needs.

There is little to no guidance in trauma-focused therapy protocols to address clinical complexities and modify therapy accordingly. The perception of a forced choice between 1.) adherence to a manualized therapy and 2.) personalizing the protocol to best meet the patient's needs, leads to higher levels of dropout and poorer outcomes. Overly rigid adherence to the treatment protocol is a common contributor to CPT dropout. In the face of treatment challenges, one-half of patients received a modified trauma-focused therapy. However, patients who completed modified trauma-focused treatment had significantly worse outcomes than Veterans who completed standard trauma-focused therapy. The rationale for and content of the modifications was unknown. The other half of complex cases were switched to a different type of therapy and PTSD was no longer the target of treatment. When faced with clinical complexities, there is no guidance for therapists to expand and enhance the protocol to accommodate patient needs, leaving therapists to initiate strategies lacking in evidence or abandon treating PTSD altogether to target the clinical complexity.

Integrating a case formulation (CF) approach into the existing CPT protocol will enable providers to simultaneously address Veterans' clinical complexities that interfere with CPT delivery and enhance functional outcomes, while maintaining fidelity to effective CPT principles. CF is a patient-centered, collaborative process between providers and patients. CF allows providers to tailor cognitive-behavioral treatments to specific patients' unique clinical complexities within clear parameters of what justifies divergence from the standard protocol. Integrating a case formulation approach into CPT provides therapists with the tools to effectively navigate the fine line between maintaining the trauma-focus necessary to treat PTSD and attending to the clinical complexities and functional impairments that contribute to suboptimal doses of therapy and/or poorer outcomes. This study seeks to improve the clinical effectiveness of CPT by integrating a CF approach that will enable providers to directly target impairments in functioning and flexibly address clinical complexities that arise during the delivery of the CPT protocol.

Methods To accomplish the study aims, this randomized controlled trial will utilize a national sample of VHA CPT providers. This study will increase the external validity of the project by including: (a) broad provider and Veteran inclusion criteria, (b) using field-based providers, (c) employing CPT delivered in accordance with VHA's CPT Dissemination Initiative as the comparison condition, (d) avoiding the use of study-team strategies to improve Veterans' engagement, and (e) utilizing ITT analyses. A national sample of CPT providers (n = 50) will be randomized to deliver either CPT or CF-CPT. Each provider will deliver the treatment to 4 consecutive Veterans presenting for CPT treatment in his/her clinic who consent to study participation (n=200 Veterans. Key features of this pragmatic design include substituting centralized study processes and reliance on the existing network of CPT providers instead of relying on recruitment sites and local site investigators. Methods will include (1) centralized recruitment, enrollment, & data collection, (2) enrollment & consent of study providers, and (3) consent of Veteran participants by phone with a waiver of documentation of informed consent.

Description of Treatments. Cognitive Processing Therapy: CPT is a brief therapy for PTSD predominantly based on cognitive theory. Traditionally delivered over 12 one-hour sessions weekly or twice weekly, CPT is now variable length depending on patient's recovery from PTSD. CPT is delivered in three phases: education, processing, and challenging and focuses on challenging beliefs and assumptions related to the trauma, oneself, and the world. Changing dysfunctional beliefs alters negative emotions emanating from those beliefs.

Case Formulation + CPT (CF+CPT): The CF approach builds on the success of CPT in reducing core PTSD symptoms and alters the protocol in two important ways: expanding the protocol to intentionally and systematically address impairment in functioning, and enhancing the providers' latitude to navigate challenges to optimal therapy outcomes (COTOS) that threaten patient engagement. CPT protocol expansion will occur for all patients, intentionally increasing the focus of the intervention to explicitly assess, track and intervene with impairments in functioning (Criterion G of PTSD). To accomplish this, CF-CPT begins with a formal CF assessment session; elements of CF are then integrated throughout CPT. CF modifications to the original CPT protocol occur in each session by intentionally attending to cognitions that are impeding the patient's functional recovery. The goal of the case formulation approach to CPT is to provide guidance to the therapist in increasing the patient's active involvement in CPT and personalizing the approach to best meet the patient's needs while ensuring that the trauma-focused work is prioritized.

The second modification to the original CPT protocol includes enhancing the provider's latitude to diverge from the protocol when clinically wise. The clinical complexities commonly observed during care delivery and identified as risk factors in empirical research present challenges to optimal therapy outcomes (COTOs) during recovery from PTSD. COTOs constitute any and all potential patient-level challenges or clinical issues that might arise during therapy and present obstacles to standardized administration of a manualized therapy protocol such as CPT. COTOs are central to functional outcomes and, as such, present risks to holistic recovery insofar as they 1.) increase the likelihood of premature drop-out resulting in inadequate doses of treatment, and 2.) are often considered outside the scope of trauma-focused treatment and are subsequently left unattended. The universe of possible COTOs cannot be quantified in any single protocol as they are idiosyncratic to the patient, but they can be categorized into five larger domains for ease of assessment: 1) emotional dysregulation, 2) significant avoidance behaviors 3) ambivalence and beliefs about therapy, 4) comorbid conditions, and 5) significant psychosocial and environmental stressors and crises.

Intentional assessment of these domains and identification of COTOs provides the opportunity to monitor and address the COTO before the protocol is irreparably ruptured or abandoned. As COTOs present themselves during the protocol-driven delivery of CPT, therapists face multiple decision points. In weighing competing patient needs, therapists struggle with balancing fidelity to the treatment manual and simultaneously ensuring that the patient's multifaceted needs are met. As with other single disorder protocols, CPT offers little guidance for navigating existing and emerging COTOs during treatment. By default, the global recommendation for clinicians is to stay on CPT protocol and maintain the focus on PTSD or administer a different treatment. However, too much rigidity negatively impacts patient engagement and modifications to the protocol have significantly enhanced CPT effectiveness and are now considered the standard of care. CF-CPT thus provides guidance around the identification, monitoring and management of COTOs, and, importantly, the expedient return to the CPT protocol with continued attention to the patient's idiosyncratic COTOs.

Aim 1 Methodology: Compare the effectiveness of CF-CPT as compared to CPT in improving Veterans' functioning and quality of life.

Provider Inclusion / Exclusion Criteria. Providers will include up to 56 licensed VHA clinicians who have been trained in CPT, are listed on the CPT National Provider Roster, and who self-report administering CPT to at least 7 Veterans during the prior twelve months.

Provider Recruitment. Provider recruitment and participation will occur nationally over 4 waves. From the pool of interested providers, a random, stratified sampling frame of providers who meet inclusion criteria will be developed. Stratification will include oversampling for providers who engage female patients to have an adequate representation of both genders and will be stratified by VISN to increase the likelihood that the study sample will be representative of the racial/ethnicity diversity of Veterans with PTSD nationwide. Using phased provider recruitment will enable enrollment of providers and patients at a manageable rate, adequately staff the study, and begin participation as soon after provider recruitment and training as possible to reduce the chances of therapist attrition Provider Randomization. Using a 1:1 allocation ratio, a computer-generated randomization sequence will randomize eligible providers to each study condition. Randomization will be blocked within recruitment wave. Providers will only be delivering the therapy in the condition to which they have been randomized. This will minimize therapist drift and possible contamination effects.

Veteran Inclusion / Exclusion Criteria and Recruitment. Each of the 50 providers will treat 4 CPT patients (total sample = 200) with either CF-CPT (n = 100) or CPT (n = 100), as dictated by provider randomization. To avoid selection bias in patient population, all consecutive Veterans with whom the provider is intending to begin a course of individually-delivered CPT will be offered study participation until 4 Veterans are enrolled. Thus, in order to be invited to participate, Veterans will have been identified as PTSD positive per clinic screening processes. Once Veterans express interest in participation to the CPT provider, they will complete a diagnostic interview with study staff blinded to condition in order to confirm a full diagnosis of PTSD. Study exclusion criteria include active suicidal ideation with intent, homicidality, current mania, psychosis, or serious drug or alcohol abuse that requires immediate medical attention (e.g. inpatient care). Patients should not be participating in another trauma-focused therapy at the time of enrollment but can continue any psychiatric medications (dose must be stable for one month prior to enrollment). Medication changes will not be prohibited for Veterans in either treatment arm following baseline assessment and randomization.

Study Procedures and Data Collection. Patient participants will be assessed prior to treatment (pretreatment), mid-treatment (after session 6 or 6 weeks post-randomization for treatment dropouts), 2 weeks post- treatment or 14 weeks after study initiation for treatment dropouts (posttreatment), and 12 weeks after the posttreatment assessment (follow-up). Over the course of the study, patient data will be collected by a) interviews delivered via phone, b) mailed paper and pencil survey, and c) retrieval from EMR. Veterans will complete the phone interview and survey at each assessment interval (pre, mid, post, and follow-up) and will be paid for each completed interview and for each completed packet of questionnaires.

Phone Interviews. All diagnostic clinical interviews will be conducted by an independent evaluator (IE), blinded to study condition, by telephone. IEs participate in four stages of training: relevant readings, expert-led classroom instruction, mock interviews with national experts, and co-rating exercises with previously taped assessments. After training, all IEs will engage in weekly calibration exercises to ensure maintenance of high quality standards and prevent drift in scoring.

Self-report surveys. Self-report measures will be collected at all assessment intervals online via Qualtrics or by paper and pencil. Depending on participant preference.

Measures. In addition to outcomes specified in the study specific aims, the investigators will measure constructs and conditions associated with each COTO domain. While not able to formally assess the universe of possible COTOs for each participant, the investigators selected standardized measures for those believed are most likely to arise. For those randomized to CF-CPT, the investigators will also utilize the Daily Monitoring Diary completed throughout the course of treatment as an idiosyncratic measure of all relevant COTOs for the individual patient.

Treatment Delivery. All treatment will be delivered in in-person individual therapy sessions by rostered CPT providers and will be audio-recorded.

Delivery of CPT. Providers randomized to the CPT intervention will be asked to continue to deliver the treatment in accordance with the CPT manual.

Delivery of CF-CPT. The CPT protocols will be modified with the CF-CPT approach in three ways. First CF-CPT will begin with the case formulation assessment. Feedback from the case formulation session will be incorporated into the traditional CPT session 1, allowing time to continue developing the individualized monitoring tool (daily diary). Second, patients in CF-CPT will monitor identified COTOs throughout therapy via the daily diary. Third, patients in CF-CPT will also be instructed to apply CPT specific skills to COTOs and functioning related cognitions during practice assignments, etc. Some portion of the CF-CPT group's identified COTOs will increase during the course of CPT. For only those patients for whom it is necessary, the content of the therapy may be altered accordingly.

Clinical Case Consultation and Fidelity Assessments. To ensure that each condition is delivered in the way in which it was intended, case consultation will be provided to all providers on a weekly basis. Adherence and competence will be determined by independent and expert raters who are not otherwise involved in the project.

Power Analysis. Power calculations based on mixed model tests for two means in a two-level hierarchical design with level-2 randomization to intervention group confirmed that the proposed sample (200 Veterans) adequately powers the study to detect meaningful between group differences. With an estimated sample size of 200, the study would have 83% power to detect an 8-point difference (d = 0.47) on the total IPF score.

Data Analysis: Analyses will follow ITT methodology. The investigators will test Aim 1 hypotheses using generalized linear mixed models. Continuous patient Aim 1A & 1B outcome measures (all but treatment completion), within the assumed and appropriate fitted distributions, will be modeled with treatment and training wave as fixed effects and a random provider effect (clustering by provider). The time (pretreatment, mid-treatment posttreatment, three-month follow-up) by treatment interaction term will provide the test of the investigators' primary hypothesis that CF-CPT will be superior as compared to CPT.

For the dichotomous measure of treatment completion (Aim 2), logistic mixed models with a random provider effect will be used. Given that the amount of divergence from the CPT protocol will vary across patients, the investigators will augment the primary analysis with secondary analyses comparing subsamples of the CF-CPT group (e.g., those with and without divergences) to the CPT group. This secondary analysis will require adjustments for possible covariate imbalance, as the investigators will lose the balance induced by randomization. The investigators will use propensity analysis and will estimate average treatment effect on the treated (ATT) and the corresponding sensitivity analysis to gain more insight on the magnitude of the effect. Post hoc power will also be calculated to assess the generalizability of these estimates.

Finally, the investigators will examine the COTO reduction score as a predictor of improvements in functioning and symptoms - i.e., testing whether more improvement in COTO scores is associated with greater improvement in study outcomes (Aim 3). The investigators propose adapting an idiosyncratic method of assessment via locally constructed diaries used in previous studies to track PTSD symptoms to monitor idiosyncratic COTOs and provide data to evaluate the effectiveness of the CF intervention on the individual challenges in patients' lives by calculating a Composite Primary COTO Reduction (CPCR) score. This score is an index of overall change in COTO level and can be conceptualized as a percentage of improvement. The CPCR score also provides a means for describing clinically significant improvement in symptomatology, functioning, etc.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with posttraumatic stress disorder (PTSD)

Exclusion Criteria:

* Study exclusion criteria include active suicidal ideation with intent, homicidality, current mania, psychosis, or serious drug or alcohol abuse that requires immediate medical attention (e.g. inpatient care)
* Patients should not be participating in another trauma-focused therapy at the time of enrollment but can continue any psychiatric medications (dose must be stable for one month prior to enrollment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Inventory of Psychosocial Functioning (assessing change over time) | Assesses functioning over the 30 days prior to baseline assessment, change between baseline and session 6, change over following treatment (post-treatment), and at the 3-month follow-up interval.
  This standardized self-report instrument assesses PTSD-related psychosocial functioning. The IPF is an 80-item self-report questionnaire of functional impairment across several domains including relationships, work, parenting, education, and general daily functioning over the past 30 days. Domain scores can range from 0 to 100 with higher values corresponding to higher functioning. Overall functioning score was calculated as the mean of all completed IPF domain scores. As participants may skip certain domains that do not apply to them (thus leading to different sample sizes for analyses predicting different domains of functioning), overall score was calculated as total sum of all completed IPF domain scores divided by the actual number of domains completed by the participant.
Clinician-Administered PTSD Scale-5 (CAPS) (assessing change over time) | Administered at baseline, mid-treatment (after session 6), two weeks following treatment (post-treatment), and at the 3-month follow-up interval.
  The CAPS is a 30-item structured interview that corresponds to the DSM-5 criteria for PTSD. The CAPS will be used to make a current (past month) and lifetime diagnosis of PTSD. In addition to assessing the 20 PTSD symptoms, questions target the impact of symptoms on social and occupational functioning, improvement in symptoms since a previous CAPS administration, overall response validity, overall PTSD severity, and frequency and intensity of five associated symptoms. For each item, standardized questions and probes are provided.
  CAPS-5 diagnosis demonstrated strong interrater reliability, and test-retest reliability, as well as strong correspondence with a diagnosis based on the CAPS for DSM-IV. CAPS-5 total severity score demonstrated high internal consistency, and interrater reliability, and good test-retest reliability, and good discriminant validity with measures of anxiety, depression, somatization, functional impairment, psychopathy, and alcohol abuse.

SECONDARY OUTCOMES:
WHO - Disability Assessment Schedule 2.0 (WHODAS-II) (assessing change over time) | Administered at baseline, mid-treatment (after session 6), two weeks following treatment (post-treatment), and at the 3-month follow-up interval.
  This widely used self-report questionnaire asks about difficulties experienced in relation to health conditions in six domains: understanding and communicating, getting around, self-care, getting along with people, life activities (work/school), and participation in society. The WHODAS-II has been shown to have high internal consistency, stable factor structure, and high test-retest reliability. Rigorous tests performed during the WHODAS-II development demonstrate its usability across cultures, sexes, and age groups and for a variety of diseases and health conditions. WHODAS-II was specifically developed to measure clinical outcomes and treatment effectiveness over time. It has established sensitivity to symptom change across a wide range of clinical conditions including depression and anxiety disorders, physical illness, and traumatic brain injury.
WHO - Quality of Life - Brief (assessing change over time) | Administered at baseline, mid-treatment (after session 6), two weeks following treatment (post-treatment), and at the 3-month follow-up interval.
  The World Health Organization Quality of Life - BREF (WHOQOL-BREF) is a self-report questionnaire which assesses 4 domains of quality of life (QOL): physical health, psychological health, social relationships, and environment. In addition, there are 2 items that measure overall QOL and general health. The assessment conceptually fits with the WHO definition of QOL. WHOQOL-BREF can provide data for both research and clinical purposes. Although it is a relatively brief instrument, its structure allows one to acquire specific information covering many aspects of life.
  Subscales (domains): Physical Health (7 items) Psychological Health (6 items) Social Relationships (3 items) Environment (8 items)
  Scoring: Items scored 1-5. Raw domain score is the sum of respective item scores. All domain scores are then normalized to a range of 0-100. Refer to user manual for scoring algorithm. SPSS algorithm available for automatic scoring.
Well-Being Inventory (WBI) (assessing change over time) | Administered at baseline, mid-treatment (after session 6), two weeks following treatment (post-treatment), and at the 3-month follow-up interval.
  The WBI is a multidimensional instrument that was designed to assess status, functioning, and satisfaction with four key life domains of vocation, finances, health, and social relationships. In total, there are 21 sections of the WBI and 126 questions/statements: 34 items for vocation, 24 for finances, 20 for health, and 48 for social relationships. Throughout the inventory, respondents are instructed to provide responses to categorical items (e.g., yes, no), or to endorse a single response from among statements using a 5-point Likert type response format (e.g., 1 = Never to 5 = Most or all of the time; 1 = Very dissatisfied to 5 = Very satisfied). Measures within each domain may be extracted from the full inventory and are available to use as separate entities depending on the needs of the administrator and/or the purpose of the assessment.
PTSD Checklist-DSM-5 (PCL-5) (assessing change over time) | Administered at baseline, weekly (during treatment) mid-treatment (after session 6), two weeks following treatment (post-treatment), and at the 3-month follow-up interval.
  The PCL-5 will also be used to assess PTSD. The DSM 5 civilian version was chosen because it is open to any trauma, not just combat trauma. The PCL-5 is a 20-item self-report measure of PTSD. The items correspond to the DSM-5 symptoms for PTSD and yield a total score and four symptom cluster subscale scores. Higher scores indicate more severe PTSD symptoms with scores above the clinical cutoff of 32 indicating a likely diagnosis of PTSD. The PCL-5 has excellent internal consistency, reliability and validity.
Patient Health Questionnaire - 9 (assessing change over time) | Administered at baseline, weekly (during treatment), mid-treatment (after session 6), two weeks following treatment (post-treatment), and at the 3-month follow-up interval.
  The PHQ-9 is the 9-question depression scale of the PHQ aimed to detect the severity of depression. The PHQ is a version of the PRIME-MD, a screening tool that assesses 12 mental and emotional health disorders. The PHQ is a 59-question instrument with modules on mood (PHQ-9), anxiety, alcohol, eating, and somatoform disorders. A 4-point Likert scale, ranging from 0 (not at all) to 3 (almost all of the days), is used for each item. The total score for the nine questions is added up and can range from 0 to 27. A score of greater tan 20 indicates major depression (severe), 15 and 19 indicates major depression (moderately severe), 10 to 14 indicates minor depression, dysthymia, and major depression (mild), and 5 to 9 indicates mild symptoms of depression.
session progress notes (assessing change over time) | Session progress notes will be written by clinician following each weekly treatment session through study completion (an average of three months). This will reflect participant change and progress over the course of the week as well as current status.
  Session progress notes will be gathered from patients medical records and will provide a measure of session content and therapy completion.
DSM-5 Cross-cutting symptom measure (CCSM) (assessing change over time) | Administered at baseline, mid-treatment (after session 6), and two weeks following treatment (post-treatment).
  This measure assesses comorbid mental health conditions. The CCSM consists of 23 questions in a self-report format that evaluates mental health domains that are significant across psychiatric diagnoses. It is quick and easy to administer, taking patients around 5 minutes to complete in the waiting room. There are 13 psychiatric domains in this measure: depression, anger, mania, anxiety, somatic symptoms, suicidal ideation, psychosis, sleep problems, memory, repetitive thoughts and behaviors, dissociation, personality functioning, and substance use. A 5-point scale (0-4) is used to record responses and reflect how much or how often the person has been concerned by a specific symptom over the previous 2 weeks. Additional inquiry is recommended if an individual scores a mild or slight rating, depending on the psychiatric symptom being investigated. This measure has good test-retest reliability in research settings and is useful and feasible in clinical practice.
Weekly stress inventory (assessing change over time) | Administered at baseline, mid-treatment (after session 6), and two weeks following treatment (post-treatment).
  This inventory measures minor life events and hassles. The WSI is an 87-item self-report scale used to assess the occurrence of minor stressors over a week's time. Individuals rank items on an 8-point Likert scale, with values ranging from 0 (did not occur) to 7 (extremely stressful). Two scores are obtained, the event score (WSI-E) which is the total number of events endorsed and the impact score (WSI-I), which is the summation of the subjective ratings of distress for the items endorsed.
Veterans Rand Short Form (assessing change over time) | Administered at baseline, mid-treatment (after session 6), and two weeks following treatment (post-treatment).
  This measure assesses health conditions and concerns about health conditions. The Veterans RAND 12 Item Health Survey (VR-12) is a brief, generic, multi-use, self-administered health survey comprised of 12 items. The instrument is primarily used to measure health related quality of life, to estimate disease burden and to evaluate disease-specific benchmarks with other populations. The 12 items in the questionnaire correspond to eight principal physical and mental health domains including general health perceptions; physical functioning; role limitations due to physical and emotional problems; bodily pain; energy-fatigue, social functioning and mental health.. The 12 items are summarized into two scores, a "Physical Health Summary Measure {PCS-physical component score}" and a "Mental Health Summary Measure {MCS-mental component score}". These provide an important contrast between physical and psychological health status.
Pittsburgh Sleep Quality Index (PSQI) (assessing change over time) | Administered at baseline, mid-treatment (after session 6), and two weeks following treatment (post-treatment).
  This measure assesses the presence and severity of several indices of sleep quality. A nineteen item survey measures assesses sleep quality. The scale yields a total score (seven component scores summed) with clinical cutoffs of scores greater than 5 indicating significant sleep disturbance. A score of greater than 5 yields diagnostic sensitivity of 89% and specificity of 86%.
PEG measure (assessing change over time) | Administered at baseline, mid-treatment (after session 6), and two weeks following treatment (post-treatment).
  This measure assesses chronic pain. The PEG is an ultra-brief measure of pain (derived from the Brief Pain Inventory). The PEG score is the average of the 3 individual item scores. Item 1 uses a Likert scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine). Items 2 and 3 use a Likert scale ranging from 0 (does not interfere) to 10 (completely interferes). For clinical use, round to the nearest whole number.
State-Trait Anxiety Inventory (assessing change over time) | Administered at baseline, mid-treatment (after session 6), and two weeks following treatment (post-treatment).
  This measure assesses severity of state anxiety (situational) and trait anxiety (enduring). The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. Range of scores for each subtest is 20-80, the higher score indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms for the S-Anxiety scale; however, other studies have suggested a higher cut score of 54-55 for older adults.
Emotional Reactivity and Numbing Scale (assessing change over time) | Administered at baseline, mid-treatment (after session 6), and two weeks following treatment (post-treatment).
  This scale assesses affective arousal across the spectrum of aroused and agitated to devoid of emotion and numb. The Emotional Numbing and Re-activity Scale is a self-report measure designed to assess the withdrawal of awareness of emotional responses to events or experiences. 36 items were administered assessing General Numbing (8 items), as well as numbing of the specific emotions of Fear (6 items), Sadness (12 items), and Anger (10 items). Each item is rated on a 5-point Likert-type scale ranging from 1= not at all typical of me to 5=entirely typical of me.
Dimensions of Anger Reactions (assessing change over time) | Administered at baseline, mid-treatment (after session 6), and two weeks following treatment (post-treatment).
  This measure assesses angry reactions/reactivity. The Dimensions of Anger Reactions scale (DAR-5) is a 5-item assessment of recent anger reactions using a 5-point Likert scale from 1 (none or almost none of the time) to 5 (all or almost all of the time). Internal consistency reliability was good for this scale, 0.91.
Beck Suicidal Ideation Scale (assessing change over time) | Administered at baseline, mid-treatment (after session 6), and two weeks following treatment (post-treatment).
  This measure assesses suicidal ideation. This scale is a 19-items instrument that evaluates the presence and intensity of suicidal thoughts in a week before evaluation. Self-reporting edition of the scale was introduced in 1988. Each item is scored based on an ordinal scale from 0 to 2 and the total score is 0 to 38. Individuals answer to the first 5 items which is excerpted. If individual's answer to the fifth item is positive (scores 1 and 2), he/she answers the rest of the items and otherwise the questionnaire is completed.
Brief Addiction Monitor (assessing change over time) | Administered at baseline, mid-treatment (after session 6), and two weeks following treatment (post-treatment).
  This measure assesses alcohol and drug use and craving. The Brief Addiction Monitor (BAM) is a 17-item, multidimensional, progress-monitoring instrument for patients in treatment for a substance use disorder (SUD). The BAM includes items that assess risk factors for substance use, protective factors that support sobriety, and drug and alcohol use (items 4-7G). The BAM produces composite scores for the three aforementioned domains. The instrument can be used in treatment planning, progress monitoring, and group or individual psychotherapies for SUD.
University of Rhode Island Change Assessment (assessing change over time) | Administered at baseline, mid-treatment (after session 6), and two weeks following treatment (post-treatment).
  University of Rhode Island Change Assessment is a widely-used 32-item self-report measure of RTC, which assesses four stages of change (pre-contemplation, contemplation, preparation/action, and maintenance). The factor structure was validated in two outpatient samples and each subscale had good internal consistency (a's = .88 to .89). Items are rated on a 5-point Likert-type scale from 1 (strongly disagree) to 5 (strongly agree) and averaged within subscales to create subscale scores. A composite readiness scale also includes cutoffs to produce a stage of change based on the total readiness score, which was used only for descriptive purposes in the current study. The current study utilized the original form of the URICA with specific instructions to focus on "trauma symptoms". This procedure is in line with the majority of previous studies using MI as a precursor to CBT. Internal consistency for each subscale in the current study was high (a's = .80 to .91).
Daily monitoring diary (assessing change over time) | Administered at baseline, daily throughout therapy, and two weeks following treatment (post-treatment).
  This idiosyncratic measures assesses the frequency and severity of any challenges to optimal therapy outcomes described by the participant in the case formulation session. The diaries are locally constructed and assess challenges to optimal therapy outcomes. The frequency and intensity of each challenge is assessed daily on a 0-5 likert scale. Change over time can be calculated using a formula to derive a composite symptom reduction score. This score can be interpreted as a percent improvement over a specified timeframe.
PhenX Demographic Questionaire | Administered at baseline.
  This measure records demographic variables including age, gender, education, marital status, parental status etc.
Life Events Checklist 5 (assessing change over time) | Administered at baseline, mid-treatment (after session 6), two weeks following treatment (post-treatment), and three months following treatment. .
  The Life Events Checklist for DSM-5 (LEC-5) is a self-report measure designed to screen for potentially traumatic events in a respondent's lifetime. The LEC-5 assesses exposure to 16 events known to potentially result in PTSD or distress and includes one additional item assessing any other extraordinarily stressful event not captured in the first 16 items.
  The LEC-5 is intended to gather information about the potentially traumatic experiences a person has experienced. There is no formal scoring protocol or interpretation per se, other than identifying whether a person has experienced one or more of the events listed. Respondents indicate varying levels of exposure to each type of potentially traumatic event included on a 6-point nominal scale, and respondents may endorse multiple levels of exposure to the same trauma type. The LEC-5 does not yield a total score or composite score.
Trauma Interview | Administered at baseline
  This locally constructed interview assesses the participant's trauma history over the course of the lifetime.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Ellen Galovski, PhD MA BS, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA; Shannon M. Kehle-Forbes, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (8):
- United States (8):
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - VA Pacific Islands Health Care System, Honolulu, HI, Honolulu, Hawaii
  - Southeast Louisiana Veterans Health Care System, New Orleans, LA, New Orleans, Louisiana
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - Salem VA Medical Center, Salem, VA, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No
In accordance with VA policy, a data sharing plan is not currently in place. However, data use agreements can be crafted and approved by the IRB to share data in the future.

DOCUMENTS (1):
  • Informed Consent Form (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT04407767/ICF_001.pdf